CLINICAL TRIAL: NCT05151198
Title: A Smartphone-based Self-management Support Program for Patients With Chronic Obstructive Pulmonary Disease - A Needs Assessment Survey
Brief Title: Smartphone-based Self-management in COPD Patients: A Needs Assessment Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant professor, The University of Hong Kong
Other Study IDs: UW21-532-1
Record Dates: First submitted 2021-11-27; First posted 2021-12-09 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Self-management; Support; Smartphone-based; Digital
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COPD patients often experience multiple symptoms (e.g. dyspnea, cough, and deteriorating quality of life) and have imposed a substantial economic and social burden on health care.

The current proposal is to explore the information needs of COPD patients and to evaluate the feasibility and acceptability of a smartphone-based instant messaging self-management support program to improve the quality of life in patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the number 3 killer globally by 2020. COPD patients often experience multiple symptoms (e.g. dyspnea, cough, and deteriorating quality of life) and have imposed a substantial economic and social burden on health care.

Current policy for the prevention and management of long-term conditions focuses on efforts to prevent the onset or slow progression of disease early in the disease trajectory. This prevention paradigm has only recently been adopted for COPD. Systematic reviews have shown self-management support for patients with COPD is effective in improving health-related quality of life and in reducing hospital admissions, but the evidence comes largely from patients with moderate or severe disease and is predominantly recruited from secondary care. Simple and systematic strategies are needed to improve out-of-hospital support and management for people living with COPD.

An instant messaging smartphone app, which allows texts, audio, pictures and video messages to be shared in chat groups, is already available to and is the most popular in the Hong Kong general public. Mobile instant messaging can be conducted through a daily use device to increase access and efficacy, which has been suggested as a feasible approach to delivering an intervention with positive effects on health behaviours and outcomes. Text messaging via mobile phones has been shown to be effective in helping promote lifestyle change in diabetes self-management, weight loss, physical activity, smoking cessation and medication adherence with quantitative and qualitative evidence. However, we have not found messaging intervention that was applied in people with COPD, except an ongoing study of using instant text message support for patients with chronic respiratory and cardiovascular diseases.

Hence, the current proposal is to use a quantitative survey and qualitative interview exploring the information needs of COPD patients and evaluating the feasibility and acceptability of a smartphone-based instant messaging self-management support program to improve the quality of life in patients with COPD.

ELIGIBILITY:
Inclusion criteria

* Aged 18 years and above
* Diagnosis with COPD
* Able to speak and read Chinese
* Able to complete the self-administered questionnaire
* Mental, cognitive and physically fit determined by the clinician or responsible investigator
* Signed informed consent

Exclusion criteria

* Serious active infection
* Severe respiratory insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Information and support needs | Baseline
  Information preferences and needs of support measured by outcome-based questions

SECONDARY OUTCOMES:
Patient Activation | Baseline
  Knowledge, skills and confidence in self-management measured by a 13-item Patient Activation Measure
Technological literacy | Baseline
  Knowledge and confidence in using instant messaging measured by outcome-based questions
Attitude towards smartphone-based intervention | Baseline
  Attitude towards smartphone-based intervention measured by outcome-based questions

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Need to obtain consent from patients before agreeing to share individual participants data.
Supporting Information: Study Protocol
Time Frame: When study finished
Access Criteria: The minimal anonymized dataset will be available upon request to interested researchers. For interested researchers, please contact, Ms Asa Choi (email asachoi@hku.hk), (School of Nursing, The University of Hong Kong) for further information.

REFERENCES:
- [Background] Buttery SC, Zysman M, Vikjord SAA, Hopkinson NS, Jenkins C, Vanfleteren LEGW. Contemporary perspectives in COPD: Patient burden, the role of gender and trajectories of multimorbidity. Respirology. 2021 May;26(5):419-441. doi: 10.1111/resp.14032. Epub 2021 Mar 9. PMID 33751727
- [Background] Jolly K, Sidhu MS, Hewitt CA, Coventry PA, Daley A, Jordan R, Heneghan C, Singh S, Ives N, Adab P, Jowett S, Varghese J, Nunan D, Ahmed K, Dowson L, Fitzmaurice D. Self management of patients with mild COPD in primary care: randomised controlled trial. BMJ. 2018 Jun 13;361:k2241. doi: 10.1136/bmj.k2241. PMID 29899047
- [Background] Hall AK, Cole-Lewis H, Bernhardt JM. Mobile text messaging for health: a systematic review of reviews. Annu Rev Public Health. 2015 Mar 18;36:393-415. doi: 10.1146/annurev-publhealth-031914-122855. PMID 25785892
- [Background] Redfern J, Hyun K, Singleton A, Hafiz N, Raeside R, Spencer L, Carr B, Caterson I, Cullen J, Ferry C, Santo K, Hayes A, Leung RWM, Raadsma S, Swinbourne J, Cho JG, King M, Roberts M, Kok C, Jenkins C, Chow C. ITM support for patients with chronic respiratory and cardiovascular diseases: a protocol for a randomised controlled trial. BMJ Open. 2019 Mar 1;9(3):e023863. doi: 10.1136/bmjopen-2018-023863. PMID 30826759
- See also: The top 10 causes of death — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death